CLINICAL TRIAL: NCT05540080
Title: Simultaneous Application of High-Intensity Focused Electromagnetic Procedure and Radiofrequency for Non-invasive Lipolysis and Improvement of Muscle Tone in Lateral Abdomen
Brief Title: Non-invasive Lipolysis and Improvement of Muscle Tone in Lateral Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899_CTUS700
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Fat Burn
Keywords: muscle toning; fat reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Evaluation of change in adipose and muscle layer thickness (Experimental): Evaluation of change in adipose and muscle layer thickness between pre-treatment and post-treatment based on MRI imaging and waist circumference measurements
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — Treatment with applicators C4/C5 to the BTL-899 system.

SUMMARY:
This study will evaluate the clinical efficacy and performance of the BTL-899 device for changes in subcutaneous fat and muscle tissue in the lateral abdomen region (also referred to as flanks or "love handles"). The study is a prospective, multi-center, open-label, single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and two follow-up visits. All of the study subjects will receive the treatment with the subject device.

DETAILED DESCRIPTION:
At the baseline visit, MRI imaging will be performed; the subject's weight and waist circumference will be recorded. Digital photographs of the treated area will be taken.

The treatment administration phase will consist of four (4) treatments, delivered 5-10 days apart. The applicators of BTL-899 will be applied over the area of flanks. The device will induce visible muscle contractions along with heating of the subcutaneous fat. Each therapy session will last 30 minutes.

At the last therapy visit, the subject's weight and waist circumference will be recorded, and digital photographs of the treated area will be taken. In addition, subjects will receive Therapy Comfort and Subject Satisfaction Questionnaire to fill in.

Safety measures will include documentation of adverse events (AE), which will be assessed after each procedure and at all of the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 years and older
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain their regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* A metal-containing intrauterine device (IUD)
* Swollen or neoplastic tissues, space-occupying lesions or skin eruptions in the treatment area
* Graves' disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in adipose and muscle layer thickness | 4 months
  The changes in muscles and adipose tissue of the treatment area between pre-treatment and post-treatment will be evaluated according to the MRI imaging and waist circumference measurements.
  Using the obtained MRI images, changes in adipose and muscular tissues before and after the therapy sessions will be compared for every participant according to the study phase.
  The circumference before and after the study therapy will be compared for each subject, according to the study phase. The circumference will be measured to identify any change in abdominal circumference related to changes in adipose tissue and muscle thickness.
  When applicable, the statistical analysis will be conducted in Microsoft Excel spreadsheet software with a level of significance set to 5%.

SECONDARY OUTCOMES:
Subject Satisfaction | 4 months
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for an analysis of the subject's opinion of the therapy results, where the best possible answer would be "strongly agree" and the worst "strongly disagree".

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Georgia Plastic & Reconstructive Surgery, Marietta, Georgia
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois
  - New Jersey Plastic Surgery (NJPS), Montclair, New Jersey
  - Integrated Aesthetics, Spring, Texas

IPD SHARING:
Plan to Share IPD: No